CLINICAL TRIAL: NCT02077465
Title: A Phase 1 Double-Blind, Randomized, Placebo-Controlled, Multicenter Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GS-5745 in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Safety, Tolerability, and Pharmacokinetics of Andecaliximab in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-368-1212
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, chronic obstructive pulmonary disease; Safety, Pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — andecaliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Andecaliximab (Experimental): Participants will receive andecaliximab every 2 weeks for a total of 3 infusions.
  Interventions: Drug: Andecaliximab
- Placebo to match andecaliximab (Placebo Comparator): Participants will receive placebo to match andecaliximab every 2 weeks for a total of 3 infusions.
  Interventions: Drug: Placebo to match Andecaliximab

INTERVENTIONS:
Drug: Andecaliximab — 400 mg andecaliximab administered intravenously
  Other Names: GS-5745
  Arms: Andecaliximab
Drug: Placebo to match Andecaliximab — Placebo to match andecaliximab administered intravenously
  Arms: Placebo to match andecaliximab

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of multiple infusions of andecaliximab (formerly GS-5745) in participants with chronic obstructive pulmonary disease (COPD) as assessed by adverse events (AEs) and laboratory abnormalities.

ELIGIBILITY:
Key Inclusion Criteria:

* Weight: ≥ 45 kg to < 120 kg at screening
* Males or non-pregnant, non-lactating females
* Male individuals and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception. Male individuals must refrain from sperm donation for 90 days post last infusion of the study drug
* Diagnosis of COPD per Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines for at least 6 months prior to screening and anticipated to remain on stable therapy for the duration of the study
* Post-bronchodilator forced expiratory volume in one second (FEV1) ≥ 40% predicted
* No changes in COPD medications within 30 days prior to randomization
* Hepatic panel [aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, direct bilirubin, alkaline phosphatase, lactate dehydrogenase (LDH)] ≤ 2 times the upper limit of the normal range (ULN)
* Serum creatinine ≤ 2.0
* Hemoglobin ≥ 8.5 g/dL (both males and females)
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1,500 mm^3)
* Platelets ≥ 100 x 10^9/L

Key Exclusion Criteria:

* Clinically significant active infection as judged by the investigator during screening
* Known history of HIV, hepatitis B or C during screening. Individuals who are hepatitis B surface antigen positive, but who received a successful series of hepatitis B vaccinations and never had the disease remain eligible
* A positive QuantiFERON-TB GOLD test during screening
* History of malignancy within the last 5 years except for patients who have been treated locally for non-melanoma skin cancer or cervical carcinoma in situ
* Any serious cardiac event such as myocardial infarction, unstable or life-threatening arrhythmia, hospitalization for cardiac failure within 6 months prior to randomization or any significant or new electrocardiogram (ECG) finding at Visit 1 as judged by the Investigator
* A hospitalization for a respiratory event such as, but not limited to, COPD, pneumonia, bronchiolitis, within the previous 6 months prior to randomization
* Chronic lung disease other than COPD such as: asthma, cystic fibrosis or fibrotic disease, α-1-antitrypsin deficiency, interstitial lung disease, pulmonary thromboembolic disease, or bronchiectasis
* Chronic use of systemic corticosteroids and/or treatment with systemic corticosteroids for an acute exacerbation of COPD (AECOPD) event, or other medical condition not requiring hospitalization, within 90 days of randomization.
* Treatment with antibiotics for an AECOPD event, or other medical condition not requiring hospitalization within 90 days of randomization, or any minor medical event not requiring hospitalization within 14 days of randomization.
* Treatment with any marketed or investigational biologic within 5 half-lives of the molecule or if unknown within 90 days of screening
* Individuals currently on nonbiologic immune modulator medications such as: azathioprine, cyclosporine, hydroxychloroquine, leflunomide, methotrexate, mycophenolate mofetil, sulfasalazine, tofacitinib, within 90 days of randomization

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2014-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - Advanced Pharma CR, LLC, Miami, Florida
  - Elite Research Institute, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - University at Buffalo CTRC, Buffalo, New York
  - Volunteer Research Group, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 11 March 2014. The last study visit occurred on 27 October 2014.
Pre-assignment Details: 33 participants were screened.
Groups:
- Andecaliximab: Participants received intravenous (IV) infusion of andecaliximab (400 mg) once every 2 weeks for a total of 3 infusions.
- Placebo: Participants received IV infusion of placebo once every 2 weeks for a total of 3 infusions.
Period: Overall Study
Arm/Group | Andecaliximab | Placebo
Started | 8 | 3
Completed | 7 | 2
Not Completed | 1 | 1
Not completed — Withdrew Consent | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 infusion of study drug (andecaliximab or placebo).
Groups:
- Andecaliximab: Participants received IV infusion of andecaliximab 400 mg once every 2 weeks for a total of 3 infusions.
- Total: Total of all reporting groups
Arm/Group | Andecaliximab | Placebo | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (3.3) | 56 (3.5) | 62 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2 | 1 | 3
  White | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: First dose date up to Day 29 plus 30 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab | Placebo
Number analyzed (Participants) | 8 | 3
percentage of participants | 75.0 | 33.3

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from baseline and occurring after the first dose of study drug and within 30 days after last study drug administration. The severity of laboratory abnormalities was assessed as Grade 0, 1 (mild), 2 (moderate), 3 (severe), or 4 (potentially life threatening) using the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: First dose date up to Day 29 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab | Placebo
Number analyzed (Participants) | 8 | 3
percentage of participants
  Any Post-Baseline Toxicity Grade | 87.5 | 100.0
  Grade 1 | 75.0 | 100.0
  Grade 2 | 12.5 | 0.0
  Grade 3 | 0.0 | 0.0
  Grade 4 | 0.0 | 0.0

3. Primary Outcome: Percentage of Participants Who Developed Anti-andecaliximab Antibodies
Description: The presence of anti-andecaliximab antibodies in serum samples was determined using an electrochemiluminescent (ECL) assay that detects antibodies that bind to andecaliximab.
Time Frame: Day 43
Population: The immunogenicity analysis set included participants who received any amount of andecaliximab.
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab
Number analyzed (Participants) | 8
percentage of participants
  Day 43 Positive Anti-Drug Antibody (ADA) Response | 12.5
  Day 43 Negative ADA Response | 75.0
  Unknown (no ADA sample available) | 12.5

4. Secondary Outcome: Pharmacokinetic (PK) Parameter of Andecaliximab: AUClast for Days 1, 15 and 29
Description: AUClast is defined as the area under the plasma concentration versus time curve from time zero to the last quantifiable concentration. Data for Day 1 was generated based on the data collected from Day 1 through Day 15. Data for Day 15 was generated based on the data collected from Day 15 through Day 29. Data for Day 29 was generated based on the data collected from Day 29 through Day 43.
Time Frame: Day 1 (pre-infusion; 30 minutes and 4 hours post end of infusion), Day3, Day 8, Day 15 (pre-infusion; and 30 minutes post end of infusion), Day 29 (pre-infusion; and 30 minutes post end of infusion), Day 36 and Day 43; Infusion duration = 30 to 35 minutes
Population: The PK analysis set included all participants in the safety analysis set who have an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Andecaliximab
Number analyzed (Participants) | 8
day*ug/mL
  Day 1 | 1206.7 (357.75)
  Day 15 | 1880.5 (600.33)
  Day 29 | 1822.2 (283.39)

5. Secondary Outcome: PK Parameter of Andecaliximab: AUCinf for Day 1
Description: AUCinf is defined as the area under the plasma concentration versus time curve extrapolated to infinite time. Data for Day 1 was generated based on the data collected from Day 1 through Day 15.
Time Frame: Day 1 (pre-infusion; 30 minutes and 4 hours post end of infusion), Day 3, Day 8, and Day 15 (pre-infusion); Infusion duration = 30 minutes to 35 minutes
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Andecaliximab
Number analyzed (Participants) | 7
day*ug/mL | 1398.1 (265.26)

6. Secondary Outcome: PK Parameter of Andecaliximab: %AUCexp for Day 1
Description: %AUCexp is defined as the percentage of AUC extrapolated between AUClast and AUCinf. Data for Day 1 was generated based on the data collected from Day 1 through Day 15.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of AUC
Arm/Group | Andecaliximab
Number analyzed (Participants) | 7
percentage of AUC | 19.97 (12.781)

7. Secondary Outcome: PK Parameter of Andecaliximab: Cmax for Days 1, 15 and 29
Description: Cmax is defined as the maximum observed plasma concentration of drug. Data for Day 1 was generated based on the data collected from Day 1 through Day 15. Data for Day 15 was generated based on the data collected from Day 15 through Day 29. Data for Day 29 was generated based on the data collected from Day 29 through Day 43.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Andecaliximab
Number analyzed (Participants) | 8
ug/mL
  Day 1 | 236.7 (62.70)
  Day 15: number analyzed (Participants) | 6
  Day 15 | 255.9 (71.25)
  Day 29: number analyzed (Participants) | 6
  Day 29 | 270.6 (46.48)

8. Secondary Outcome: PK Parameter of Andecaliximab: Tmax for Days 1, 15 and 29
Description: Tmax is defined as the time (observed time point) of Cmax. Data for Day 1 was generated based on the data collected from Day 1 through Day 15. Data for Day 15 was generated based on the data collected from Day 15 through Day 29. Data for Day 29 was generated based on the data collected from Day 29 through Day 43.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Andecaliximab
Number analyzed (Participants) | 8
day
  Day 1 | 0.08 (0.076)
  Day 15: number analyzed (Participants) | 6
  Day 15 | 0.02 (0.000)
  Day 29: number analyzed (Participants) | 6
  Day 29 | 0.02 (0.001)

9. Secondary Outcome: PK Parameter of Andecaliximab: Clast for Days 1, 15 and 29
Description: Clast is defined as the last observable concentration of drug. Data for Day 1 was generated based on the data collected from Day 1 through Day 15. Data for Day 15 was generated based on the data collected from Day 15 through Day 29. Data for Day 29 was generated based on the data collected from Day 29 through Day 43.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Andecaliximab
Number analyzed (Participants) | 8
ug/mL
  Day 1 | 37.07 (18.740)
  Day 15: number analyzed (Participants) | 6
  Day 15 | 50.27 (14.724)
  Day 29: number analyzed (Participants) | 6
  Day 29 | 71.74 (23.905)

10. Secondary Outcome: PK Parameter of Andecaliximab: Tlast for Days 1, 15 and 29
Description: Tlast is defined as the time (observed time point) of Clast. Data for Day 1 was generated based on the data collected from Day 1 through Day 15. Data for Day 15 was generated based on the data collected from Day 15 through Day 29. Data for Day 29 was generated based on the data collected from Day 29 through Day 43.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Andecaliximab
Number analyzed (Participants) | 8
day
  Day 1 | 12.96 (2.582)
  Day 15: number analyzed (Participants) | 6
  Day 15 | 14.79 (1.737)
  Day 29: number analyzed (Participants) | 6
  Day 29 | 13.45 (1.379)

11. Secondary Outcome: PK Parameter of Andecaliximab: λz for Day 1
Description: λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug. Data for Day 1 was generated based on the data collected from Day 1 through Day 15.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/day
Arm/Group | Andecaliximab
Number analyzed (Participants) | 7
1/day | 0.137 (0.0263)

12. Secondary Outcome: PK Parameter of Andecaliximab: CL for Day 1
Description: Clearance (CL) is defined as the systemic clearance of the drug following intravenous administration. Data for Day 1 was generated based on the data collected from Day 1 through Day 15.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Andecaliximab
Number analyzed (Participants) | 7
mL/day | 296.5 (64.67)

13. Secondary Outcome: PK Parameter of Andecaliximab: Vz for Day 1
Description: Vz is defined as the volume of distribution of the drug after intravenous administration. Data for Day 1 was generated based on the data collected from Day 1 through Day 15.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Andecaliximab
Number analyzed (Participants) | 7
mL | 2200.9 (442.03)

14. Secondary Outcome: PK Parameter of Andecaliximab: Vss for Day 1
Description: Vss is defined as the volume of distribution of the drug at steady state after intravenous administration. Data for Day 1 was generated based on the data collected from Day 1 through Day 15.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Andecaliximab
Number analyzed (Participants) | 7
mL | 2178.7 (450.66)

15. Secondary Outcome: PK Parameter of Andecaliximab: t1/2 for Day 1
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug. Data for Day 1 was generated based on the data collected from Day 1 through Day 15.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Andecaliximab
Number analyzed (Participants) | 7
day | 5.24 (1.102)

ADVERSE EVENTS:
Time Frame: First dose date up to Day 29 plus 30 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 infusion of study drug (andecaliximab or placebo).
Groups:
- Andecaliximab: Participants received IV infusion of andecaliximab 200 mg once every 2 weeks for a total of 3 infusions.
Arm/Group | Andecaliximab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 6/8 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab (N=8) | Placebo (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years